CLINICAL TRIAL: NCT06952530
Title: A Master Protocol to Investigate the Efficacy and Safety of Orforglipron Once Daily in Participants With Hypertension and Obesity or Overweight: Randomized, Double-Blind, Placebo-Controlled Trials (ATTAIN-HYPERTENSION)
Brief Title: A Master Protocol Study of Orforglipron (LY3502970) in Participants With Hypertension and Obesity or Overweight (ATTAIN-Hypertension) GZL2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27360; J2A-MC-GZL2 (Other: Eli Lilly and Company); J2A-MC-GZPL (Other: Eli Lilly and Company)
Record Dates: First submitted 2025-04-21; First posted 2025-05-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — orforglipron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Orforglipron (Experimental): Participants will receive orforglipron orally.
  Interventions: Drug: Orforglipron
- Placebo (Placebo Comparator): Participants receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Orforglipron — Administered orally
  Other Names: LY3502970
  Arms: Orforglipron
Drug: Placebo — placebo administered
  Arms: Placebo

SUMMARY:
GZL2 is an independent study conducted under the GZPL master protocol. GZL2 study will evaluate the efficacy and safety of orforglipron for treatment of hypertension in participants with obesity or overweight.

ELIGIBILITY:
Inclusion Criteria:

* refer to the GZPL master protocol study for screening eligibility.

Exclusion Criteria:

* refer to the GZPL master protocol study for screening eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in office Systolic Blood Pressure (SBP) | Baseline to Week 36

SECONDARY OUTCOMES:
Change from Baseline in 24-hour Ambulatory Blood Pressure Monitoring (ABPM) SBP | Baseline to Week 36
Percent Change from Baseline in Body Weight | Baseline to Week 36
Percent Change from Baseline in Lipids Triglycerides | Baseline to Week 36
Percent Change from Baseline in Lipids non-HDL Cholesterol | Baseline to Week 36
Percent Change from Baseline in hsCRP Concentration (mg/L) | Baseline to Week 36
Percent Change from Baseline in office SBP in Randomized Withdrawal Population | Baseline to Week 36
Pharmacokinetics (PK): Steady-State Area under the Concentration Curve (AUC) of Orforglipron | Baseline to Week 36

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (100):
- United States (30):
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Valley Clinical Trials, Inc., Covina, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Care Access - Brandon, Brandon, Florida
  - Northeast Research Institute - Downtown Office, Jacksonville, Florida
  - Peace River Cardiovascular Center, Port Charlotte, Florida
  - Care Access - St. Petersburg, St. Petersburg, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - Ascension Saint Agnes Heart Care, Baltimore, Maryland
  - Lucida Clinical Trials, New Bedford, Massachusetts
  - Arcturus Healthcare , PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Excel Clinical Research, LLC, Las Vegas, Nevada
  - Palm Research Center Sunset, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - Remington-Davis, Inc, Columbus, Ohio
  - PriMED Clinical Research, Dayton, Ohio
  - Advanced Research Institute - Tigard, Tigard, Oregon
  - Care Access - Mauldin, Mauldin, South Carolina
  - Dallas Heart and Vascular Consultants, PA, Duncanville, Texas
  - Texas Institute of Cardiology, PA, McKinney, Texas
  - North Hills Family Medicine/North Hills Medical Research, North Richland Hills, Texas
  - Advanced Research Institute, Ogden, Utah
  - Carient Heart & Vascular - Manassas, Manassas, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - National Clinical Research, Inc, Richmond, Virginia
  - Eastside Research Associates, Redmond, Washington
- Argentina (8):
  - Instituto Médico Especializado (IME), Buenos Aires
  - CIPREC, Buenos Aires
  - CEMEDIC, Buenos Aires
  - Instituto de Investigaciones Clínicas Córdoba, Córdoba
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - INECO Neurociencias Oroño, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - Santa Maria de la Salud Centro Medico, San Isidro
- China (12):
  - Beijing Pinggu District Hospital, Beijing
  - China-Japan Union Hospital, Changchun
  - Changde First People's Hospital, Changde
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second Affiliated Hospital of Chongqing Medical University - Yuzhong Campus, Chongqing
  - Jinan Central Hospital, Jinan
  - Lishui Central Hospital, Lishui
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Siping Central People's Hospital, Siping
  - Wuxi People's Hospital, Wuxi
  - Shaanxi provincial people's hospital, Xi'an
- Czechia (9):
  - Top Moravia Health, Brno
  - Ordinace Rihackovi, s.r.o., Brno
  - CTC Hodonin s.r.o., Hodonín
  - MUDr. Sarka Drinkova, Ledeč nad Sázavou
  - CCR Ostrava s.r.o, Ostrava
  - Diahelp s.r.o, Pardubice V
  - Clinoxus, Prague
  - Angiocentrum Komorany, Prague
  - Praglandia s.r.o, Prague
- Germany (9):
  - Zentrum für klinische Studien Bad Homburg, Bad Homburg
  - FutureMeds GmbH, Berlin
  - Zentrum fur klinische Forschung - Köln, Cologne
  - Hausärztlich-Kardiologisches MVZ am Felsenkeller GmbH/Zentrum für klinische Studien, Dresden
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizentrum Essen Borbeck, Essen
  - AmBeNet GmbH, Leipzig
  - Familienmedizinisches Zentrum Radowsky, Leipzig
  - RED-Institut GmbH, Oldenburg
- Greece (6):
  - Athens Medical Center - Psychikon branch, Athens
  - General Hospital of Athens "G. Gennimatas", Athens
  - University Hospital of Ioannina, Ioannina
  - G. Gennimatas General Hospital of Thessaloniki, Thessaloniki
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
- India (4):
  - Life Care Hospital and Research Centre, Bangalore
  - All India Institute of Medical Sciences, Bhubaneswar
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Ashirwad Hospital and Research Centre, Ulhasnagar
- Japan (5):
  - Tokyo-Eki Center-building Clinic, Chūōku
  - Fukuwa Clinic, Chūōku
  - Takai Internal Medicine Clinic, Kamakura-shi
  - Mikannohana Clinic, Diabetes, Endocrinology and Metabolism, Matsuyama
  - Medical Corporation Yuga Tsuruma Kaneshiro Diabetes Clinic, Yamato-shi
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Centrum Medyczne "Hipokrates" S.C. Elżbieta I Grzegorz Grześk, Bydgoszcz
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - IRMED, Piotrkow Trybunalski
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - Private Practice - Dr. Robert Witek, Tarnów
  - Balsam Medica, Warsaw
  - NZOZ Regionalna Poradnia Diabetologiczna, Wroclaw
- Puerto Rico (2):
  - Dorado Medical Complex, Dorado
  - Puerto Rico Medical Research, Ponce
- Spain (7):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital San Rafael - La Coruña, A Coruña
  - EAP Sardenya, Barcelona
  - EAP Osona Sud - Alt Congost S.L.P, Centelles
  - Complejo Asistencial Universitario de León - Hospital de León, León
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
  - Hospital Quiron Infanta Luisa, Seville

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org